CLINICAL TRIAL: NCT03999593
Title: Long-term Morbidity After Surgery for Perihilar Cholangiocarcinoma; a Cohort Study
Brief Title: Long-term Morbidity After Surgery for Perihilar Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Cholangiocarcinoma; Surgery--Complications
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Resection of perihilar cholangiocarcinoma — Resection of perihilar cholangiocarcinoma

SUMMARY:
Surgery for perihilar cholangiocarcinoma offers the only possibility of long-term survival, but remains a formidable undertaking. Traditionally, 90 day post-operative complications and death have been used to define operative risk. However, there is concern that this metric may not accurately capture long-term morbidity after such complex surgery.

This is a retrospective review of a prospective database of patients undergoing surgery for perihilar cholangiocarcinoma at a Western centre between 2009-2017.

DETAILED DESCRIPTION:
Cholangiocarcinoma is an uncommon cancer, but is the second commonest primary hepatic tumour after hepatocellular carcinoma. Its incidence is rising globally with 1200 cases per year in England & Wales. Tumours may originate within the liver itself, although the majority arise at the confluence of the hepatic ducts (perihilar tumours). Surgery is the only potentially curative treatment, but remains a formidable undertaking usually requiring a major liver resection to achieve the clear surgical margins that are essential for long-term survival, followed by complex biliary reconstruction. The magnitude of this surgery is reflected in an operative mortality reported between 10-15% in most Western centres. In addition, almost half the patients suffer major complications prior to discharge from hospital.

Following such surgery, around 30-40% of patients are alive after 5 years. However, a significant minority succumb to rapid disease recurrence, with a third dying within the first year after resection. Although offering no hope of cure, systemic chemotherapy with cisplatin/gemcitabine offers a median overall survival of 11.7 months. For patients planned to undergo surgery, but found to have locally advanced and therefore irresectable disease at laparotomy, median survival with palliative chemotherapy can reach 16 months with 10% of patients alive 3 years later. It therefore seems likely that a proportion of patients undergo major surgery, at significant risk of immediate postoperative mortality or morbidity, when they may be better served by systemic chemotherapy.

Operative morbidity and mortality has traditionally been reported as death or complication occurring within the first 30 days after surgery. However, it is now clear that this 30-day cut-off underestimates the morbidity and mortality after hepatic resection with ninety-day morbidity and mortality increasingly recognised as a more appropriate measure of postoperative outcome after liver surgery. There is also a lack of evidence on the impact that contemporary enhanced recovery after surgery (ERAS) programmes may have on these outcomes.

The unique characteristics of the complex and demanding surgery required for resection of this disease means there is also a possibility of long-term complications beyond 90-days. To date, the long-term morbidity after resection has not been reported. These data are essential to allow patients to make fully informed decisions around the risks and benefits of surgery.

This study therefore aimed to characterise the long-term morbidity after resection of perihilar cholangiocarcinoma managed with an ERAS programme in a Western centre.

ELIGIBILITY:
Inclusion Criteria:

•Macroscopically complete resection of Bismuth 2-4 (peri)hilar cholangiocarcinoma with curative intent

Exclusion Criteria:

* Metastatic disease
* Failure of curative intent resection (as per operating surgeon)
* Post resection histopathological diagnosis other than cholangiocarcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing resection for perihilar cholangiocarcinoma at University Hospital Aintree between January 2009 and October 2017 were identified using a prospectively maintained database.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Perioperative morbidity | 30 day
  Clavien-Dindo complication index

SECONDARY OUTCOMES:
Perioperative morbidity | 90 day
  Clavien-Dindo complication index

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jones, Principal Investigator — University of Liverpool

IPD SHARING:
Plan to Share IPD: No